CLINICAL TRIAL: NCT06415162
Title: Evaluation of the Effects of Education on Side Effects Management and the Use of Cooling Pillowcases on Hot Flash Complaints, Sleep and Quality of Life in Women With Breast Cancer Receiving Hormone Therapy
Brief Title: Evaluation of the Effects of Using Cooling Pillowcases, on the Symptoms of Hot Flushes, Sleep and Life Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Başak Türkmen, Phd Student Internal Medicine Nursing, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriUBTURKMEN0001
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Hormone therapy; Breast cancer; Cooling pillowcase; Hot flashes; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The intervention group will fill in the 'Patient Information Form, Menopause Specific Hot Flash Scale, Pittsburgh Sleep Quality Index and FACT-B Quality of Life Scale' in the 1st week and will be given training on treatment side effects, training booklet and 'Hot Flash Diary' to record their hot flashes. The use of cooling pillowcase will be explained. In the 5th week, 'Practices for Coping with the Side Effects of Hormone Therapy Form' will be filled out to evaluate the training and the training will be repeated. In the 3rd and 7th weeks, 'Patient Follow-up Form' will be filled by telephone, and in the 5th week face to face. In the 9th week, 'Menopause Specific Hot Flush Scale, Pittsburgh Sleep Quality Index and FACT-B Quality of Life Scale' and 'Practices Form for Coping with Side Effects of Hormone Therapy' will be completed to evaluate the training given in the 5th week. The routine care and treatment of the control group will be continued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling Pillowcases (Experimental): The intervention group will be given 'Patient Information Form, Menopause Specific Hot Flash Scale, Pittsburgh Sleep Quality Index and FACT-B Quality of Life Scale' to be filled in the 1st week, training on treatment side effects, training booklet and 'Hot Flash Diary' to record the hot flashes they experience. A cooling pillowcase will be given and its use will be explained. In the 5th week, 'Practices for Coping with the Side Effects of Hormone Therapy Form' will be filled out to evaluate the training given and the training will be repeated. A total of 3 follow-ups will be carried out by using the 'Patient Follow-up Form' by telephone in the 3rd and 7th weeks and face-to-face interview in the 5th week. In the 9th week, 'Menopause Specific Hot Flush Scale, Pittsburgh Sleep Quality Index and FACT-B Quality of Life Scale' and 'Practices for Coping with Side Effects of Hormone Therapy Form' will be completed to evaluate the effectiveness of the retraining given in the 5th week.
  Interventions: Other: Cooling Pillowcases
- Control Group (No Intervention): No intervention will be given to the patients in the control group.

INTERVENTIONS:
Other: Cooling Pillowcases — No intervention will be given to the patients in the control group.
  Other Names: Control group
  Arms: Cooling Pillowcases

SUMMARY:
This study was planned to evaluate the effect of education on the management of side effects and the use of cooling pillowcase on hot flush complaints, sleep and quality of life in women with breast cancer receiving hormone therapy.

DETAILED DESCRIPTION:
It is planned to apply pre-test evaluations in the 1st week and post-test evaluations in the 9th week to the intervention (training) group consisting of women with breast cancer who agree to participate in the study. A total of 3 follow-ups will be performed on the patients in the intervention (education) group in weeks 3 and 7 by telephone interview method and in week 5 by face-to-face interview method using the Patient Follow-up Form. In addition, in order to evaluate the effectiveness of the education given to the patients in the intervention (education) group, the Practices for Coping with the Side Effects of Hormone Therapy Form will be completed in the 5th and 9th weeks.

The control group consisting of women with breast cancer who agreed to participate in the study will be administered pre-test evaluations at week 1 and post-test evaluations at week 9. The patients in the control group will not be subjected to any intervention by the researcher, their routine treatment and care will continue, and they will be followed up only once in the 5th week by phone call.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Estrogen and progesterone receptor positive, stage 1, 2, 3 or 4 primary breast cancer,
* Receiving hormone therapy (goserelin acetate subcutaneously every 4 weeks),
* Pre/Perimenopausal period,
* No sensory and emotional barriers to communication,
* Understands Turkish, can read and write,
* Patients who voluntarily agreed to participate in the study.

Exclusion Criteria:

* Receiving treatment for anxiety and/or depression,
* Receiving gabapentin treatment for neuropathic pain,
* Active viral or bacterial infection,
* Patients with a history of sleep disorders diagnosed before hormone therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Menopausal Hot Flush Scale | nine weeks
  All items in the scale are evaluated between '0' and '10' points. The highest score that can be obtained from the scale is '100' and the lowest score is '0'. The higher the score obtained from the scale, the higher the woman's level of being affected by hot flushes.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | nine weeks
  The scale consists of 7 sub-dimensions. Each of the questions including the sub-dimension is scored between 0-3. The total score of the seven sub-dimensions varies between 0-21 and gives the total score of The Pittsburgh Sleep Quality Index. A total score above 5 indicates poor sleep quality.
Functional Assessment Of Cancer Therapy-Breast (FACT-B) | nine weeks
  The responses in the scale are organised in a 5-point Likert scale where '0' means not at all, '1' means very little, '2' means a little, '3' means quite a lot and '4' means very much. Some of the statements in the scale are reversed, and while calculating the total score of the scale, the reversed statements are subtracted from four and the other statements are directly added to the scoring. The total score that can be obtained from the scale varies between 0-148. A higher total score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Turkmen, Msc., Principal Investigator — University of Health science; Semiha Akin Eroglu, Prof., Principal Investigator — University of Health science
Locations (1):
- University of Health Science, Istanbul, Turkey (Türkiye)